CLINICAL TRIAL: NCT01718938
Title: A Multicenter, Double-Blind, Randomized, Placebo- Controlled, Phase 2 Study to Evaluate Velusetrag Effects on Gastric Emptying in Subjects With Diabetic or Idiopathic Gastroparesis
Brief Title: Phase 2 Study of Velusetrag in Diabetic or Idiopathic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Collaborators: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0093
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Diabetic; Idiopathic; Delayed gastric emptying
MeSH Terms: conditions — Gastroparesis | interventions — TD-5108

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1 (Experimental): 3-way crossover of velusetrag or placebo
  Interventions: Drug: velusetrag dose 1; Drug: velusetrag dose 2; Drug: velusetrag dose 3; Drug: placebo
- Sequence 2 (Experimental): 3-way crossover of velusetrag or placebo
  Interventions: Drug: velusetrag dose 1; Drug: velusetrag dose 2; Drug: velusetrag dose 3; Drug: placebo
- Sequence 3 (Experimental): 3-way crossover of velusetrag or placebo
  Interventions: Drug: velusetrag dose 1; Drug: velusetrag dose 2; Drug: velusetrag dose 3; Drug: placebo
- Sequence 4 (Experimental): 3-way crossover of velusetrag or placebo
  Interventions: Drug: velusetrag dose 1; Drug: velusetrag dose 2; Drug: velusetrag dose 3; Drug: placebo

INTERVENTIONS:
Drug: velusetrag dose 1
  Other Names: TD-5108
Drug: velusetrag dose 2
  Other Names: TD-5108
Drug: velusetrag dose 3
  Other Names: TD-5108
Drug: placebo

SUMMARY:
This is a multicenter, randomized, double-blind, incomplete block, three period fixed sequence crossover, multicenter, placebo-controlled study. The study will assess three oral doses of velusetrag (5 mg, 15 mg, and/or 30 mg) or placebo, administered once daily in three periods of 1-week duration each, with a 1-week washout period between treatment periods, in subjects with diabetic or idiopathic gastroparesis.

Study 0093 will evaluate the effect of velusetrag in subjects with diabetic or idiopathic gastroparesis by assessing changes in gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of gastroparesis (e.g., nausea, early satiety, fullness, bloating, upper abdominal pain, retching or vomiting) for at least 3 months prior to Screening
* Body Mass Index (BMI) between 18 and 35 kg/m2, inclusive
* Gastroparesis Cardinal Symptom Index (GCSI-2W) composite score ≥2 and ≤4 at Screening
* Delayed gastric emptying, defined as a gastric emptying half-time (GE t1/2) > 160 minutes as determined by [13C]-octanoate breath test, at Screening
* Upper gastrointestinal (UGI) obstruction ruled out by endoscopy or other imaging reasonably proximal to the diagnosis of gastroparesis

Exclusion Criteria:

* Acute severe gastroenteritis within 2 weeks prior to Screening
* History of gastric outlet obstruction
* Prior history of gastric surgery, including but not limited to gastrectomy, gastric bypass, gastric banding, pyloroplasty, vagotomy, or fundoplication
* Recurrent vomiting, defined as vomiting more than 2 days per week
* Hospitalization for treatment of gastroparesis or complications of diabetes within 4 weeks prior to Screening
* Presence of thyroid dysfunction not controlled by treatment. Subjects with abnormal thyroid stimulating hormone (TSH), hypothyroidism, or hyperthyroidism at Screening
* If Type 1 or Type 2 diabetic, a glycosylated hemoglobin (HbA1c) level >10% or a glucose > 250 mg/dL at Screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Gastric emptying half time (GE t1/2) | From baseline to week 5

SECONDARY OUTCOMES:
Duration of lag time to gastric emptying (tlag) | From baseline to Week 5
Vital signs | From baseline to Day 49
  Assess the safety and tolerability in subjects with diabetic or idiopathic gastroparesis
ECGs | From baseline to Day 49
Number of adverse events | From baseline to Day 49

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Desert Sun Clinical Research, Tucson, Arizona
  - Axis Clinical Trials, Los Angeles, California
  - Ventura Clinical Trials, Ventura, California
  - Indiana University Hospital, Indianapolis, Indiana
  - GI Associates & Endoscopy Center, Jackson, Mississippi
  - Center for Digestive and Liver Diseases, Inc., Mexico, Missouri
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Northwest Gastroenterology Clinic, Portland, Oregon
  - Digestive and Liver Disease Specialists, Norfolk, Virginia

REFERENCES:
- [Derived] Kuo B, Barnes CN, Nguyen DD, Shaywitz D, Grimaldi M, Renzulli C, Canafax D, Parkman HP. Velusetrag accelerates gastric emptying in subjects with gastroparesis: a multicentre, double-blind, randomised, placebo-controlled, phase 2 study. Aliment Pharmacol Ther. 2021 May;53(10):1090-1097. doi: 10.1111/apt.16344. Epub 2021 Apr 3. PMID 33811761